CLINICAL TRIAL: NCT03163446
Title: A Multicenter, Double-Blind, Randomized, Comparative Study of the Safety, Tolerability, Efficacy, and Pharmacokinetics of CF-301 vs. Placebo in Addition to Standard-of-Care Antibacterial Therapy for the Treatment of Adult Patients With Staphylococcus Aureus Bloodstream Infections (Bacteremia) Including Endocarditis
Brief Title: Safety, Efficacy and Pharmacokinetics of CF-301 vs. Placebo in Addition to Antibacterial Therapy for Treatment of S. Aureus Bacteremia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ContraFect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF-301-102
Record Dates: First submitted 2017-05-15; First posted 2017-05-23 (Actual); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Staphylococcus Aureus Bacteremia; Staphylococcus Aureus Endocarditis
Keywords: Staphylococcus aureus; bacteremia; staphylococcal endocarditis
MeSH Terms: conditions — Staphylococcal Infections; Bacteremia | interventions — exebacase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CF-301 (Experimental): Patients will receive a single IV infusion of CF-301 in addition to standard of care (SOC) antibacterial therapy selected by the investigator.
  Interventions: Biological: CF-301
- Placebo (Placebo Comparator): Patients will receive a single IV infusion of placebo in addition to standard of care (SOC) antibacterial therapy selected by the investigator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CF-301 — CF-301, 0.25 mg/kg, given as a single 2 hour iv infusion
  Arms: CF-301
Drug: Placebo — Placebo, given as a single 2 hour iv infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy and pharmacokinetics (PK) of CF-301 in addition to background standard of care (SOC) antibacterial therapy for the treatment of Staphylococcus aureus (S. aureus) bloodstream infections (bacteremia), including endocarditis in adults. Patients will be randomized to receive a single intravenous dose of CF-301 or placebo in addition to SOC antibacterial therapy. Patients will be prescribed standard of care antibiotics selected by the investigators based on their professional experience, practice guidelines and local antibiotic susceptibility information for the treatment of S. aureus bacteremia.

CF-301 is a lysin and member of a new class of targeted protein-based antimicrobials that has demonstrated activity against S. aureus in laboratory (in vitro) and animal studies, alone and in addition to conventional antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* male or female, 18 years or older
* blood culture positive for S. aureus
* at least one sign or symptom attributable to S. aureus bacteremia
* known or suspected complicated S. aureus BSI and/or endocarditis by Modified Duke Criteria
* patient is not pregnant or breastfeeding and is not of reproductive potential or agrees to use contraception if of reproductive potential.

Exclusion Criteria:

* patient previously received CF-301.
* treatment with any potentially effective (anti-staphylococcal) systemic antibiotic for more than 72 hours within 7 days before randomization.
* presence of any removable infection source that will not be removed or debrided within 72 hours after randomization.
* brain abscess or meningitis.
* community acquired pneumonia or known polymicrobial bacteremia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (30):
  - CF-301-102 Study Site, Birmingham, Alabama
  - CF-301-102 Study Site, Sacramento, California
  - CF301-102 Study Site, Sylmar, California
  - CF-301-102 Study Site, New Haven, Connecticut
  - CF-301-102 Study Site, Newark, Delaware
  - CF-301-102 Study Site, Atlanta, Georgia
  - CF-301-102 Study Site, Augusta, Georgia
  - CF0301-102 Study Site, Decatur, Georgia
  - CF-301 Study Site, Idaho Falls, Idaho
  - CF301-102 Study Site, Chicago, Illinois
  - CF301-102 Study Site, Burlington, Massachusetts
  - CF-301-102 Study Site, Detroit, Michigan
  - CF301-102 Study Site, Royal Oak, Michigan
  - CF301-102 Study Site, St Louis, Missouri
  - CF301-102 Study site, Butte, Montana
  - CF301-102 Study Site, Omaha, Nebraska
  - CF-301-102 Study Site, Omaha, Nebraska
  - CF-301-102 Study Site, Englewood, New Jersey
  - CF301-102 Study Site, Paterson, New Jersey
  - CF-301-102 Study Site, New York, New York
  - CF-301-102 Study Site, Valhalla, New York
  - CF-301-102 Study Site, Cleveland, Ohio
  - CF301-102 Study Site, Columbus, Ohio
  - Cf-301-102, Columbus, Ohio
  - CF-301 Study Site, Toledo, Ohio
  - CF-301-102 Study Site, Bethlehem, Pennsylvania
  - Cf-301-102, Richmond, Virginia
  - CF-301-102 Study Site, Roanoke, Virginia
  - CF-301-102 Study Site, Seattle, Washington
  - CF-301-102 Study Site, Milwaukee, Wisconsin
- Belgium (5):
  - CF-301-102 Study Site #2, Brussels
  - CF301-102 Study Site, Brussels
  - CF301-102 Study Site, Edegem
  - CF301-102 Study Site, Ghent
  - CF301-102 Study Site, Leuven
- Bulgaria (2):
  - CF301-102 Study Site, Rousse
  - CF301-102 Study Site, Sofia
- Chile (2):
  - CF-301-102 Study Site, Santiago
  - CF-301-102 Study Site, Viña del Mar
- Czechia (3):
  - CF301-102 Study Site, Brno
  - CF301-102 Study Site #2, Prague
  - CF301-102 Study Site, Prague
- France (4):
  - CF301-102 Study Site, Limoges
  - CF301-102 Study Site, Lyon
  - CF301-102 Study Site, Paris
  - CF301-102 Study Site, Toulon
- Germany (4):
  - CF-301-102 Study Site #2, Berlin
  - CF-301-102 Study Site, Berlin
  - CF-301-102 Study Site, Cologne
  - CF-301-102 Study Site, Freiburg im Breisgau
- Greece (4):
  - CF301-102 Study Site #3, Athens
  - CF301-102 Study Site, Athens
  - Study Site #2, Athens
  - CF301-102 Study Site, Larissa
- Guatemala (2):
  - CF-301-102 Study Site, Guatemala City
  - CF-301-102 Study Site, Santa Rosita
- Israel (4):
  - CF301-102 Study Site, Beersheba
  - CF301-102 Study Site, Nazareth
  - CF301-102 Study Site, Safed
  - CF301-102 Study Site, Tel Litwinsky
- Italy (3):
  - CF301-102 Study Site, Bergamo
  - CF-301-102 Study Site, Busto Arsizio
  - CF-301-102 Study Site, Genoa
- Russia (4):
  - CF-301-102 Study Site, Krasnodar
  - CF-301-102 Study Site, Moscow
  - CF-301-102 Study Site, Saint Pertersburg
  - CF-301-102 Study Site #2, Saint Petersburg
- Spain (5):
  - CF-301-102 Study Site #2, Barcelona
  - Cf301-102, Barcelona
  - CF301-102 Study Site, Córdoba
  - CF301-102 Study Site, Seville
  - CF301-102 Study Site, Terrassa
- United Kingdom (5):
  - CF301-102 Study Site, Chelmsford
  - CF301-102 Study Site, Liverpool
  - CF-301-102 Study Site, London
  - CF301-102 Study Site #2, London
  - CF301-102 Study Site, Oxford

REFERENCES:
- [Derived] Fowler VG Jr, Das AF, Lipka-Diamond J, Schuch R, Pomerantz R, Jauregui-Peredo L, Bressler A, Evans D, Moran GJ, Rupp ME, Wise R, Corey GR, Zervos M, Douglas PS, Cassino C. Exebacase for patients with Staphylococcus aureus bloodstream infection and endocarditis. J Clin Invest. 2020 Jul 1;130(7):3750-3760. doi: 10.1172/JCI136577. PMID 32271718

RESULTS

PARTICIPANT FLOW:
Groups:
- CF-301: Patients received a single IV infusion of CF-301 in addition to standard of care (SOC) antibacterial therapy selected by the investigator.
- Placebo: Patients received a single IV infusion of placebo in addition to standard of care (SOC) antibacterial therapy selected by the investigator.
Period: Overall Study
Arm/Group | CF-301 | Placebo
Started | 73 | 48
Completed | 45 | 31
Not Completed | 28 | 17
Not completed — Unable to return for Day 180 visit | 2 | 0
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Death | 16 | 5
Not completed — Lost to Follow-up | 6 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Patient randomized but went to surgery and was unable to be dosed. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | CF-301 | Placebo | Total
Number analyzed (Participants) | 73 | 48 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 36 | 86
  >=65 years | 23 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (15.24) | 55.0 (15.62) | 55.9 (15.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 39
  Male | 50 | 32 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 8 | 22
  White | 51 | 30 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 58 | 38 | 96
  United Kingdom | 2 | 2 | 4
  Russia | 1 | 0 | 1
  Greece | 2 | 0 | 2
  Belgium | 1 | 1 | 2
  Guatemala | 4 | 5 | 9
  Italy | 1 | 0 | 1
  Israel | 1 | 0 | 1
  Chile | 1 | 1 | 2
  France | 1 | 0 | 1
  Germany | 1 | 1 | 2
Diagnosis [Count of Participants; unit: Participants]
  Right-sided endocarditis | 5 | 3 | 8
  Left-sided endocarditis | 10 | 3 | 13
  Right and left-sided endocarditis | 1 | 0 | 1
  Uncomplicated bloodstream infection (BSI) | 13 | 3 | 16
  Complicated bloodstream infection (BSI) | 43 | 37 | 80

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events [Safety and Tolerability]
Description: Number and percentage of patients with treatment-emergent adverse events (TEAEs)
Time Frame: Through Day 7, at Test of Cure (TOC) between 56-70 days, and at Day 180
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 72 | 47
Participants
  TEAE through Day 7 | 48 | 30
  TEAE through TOC | 64 | 40
  TEAE through Day 180 | 67 | 40

2. Primary Outcome: Clinical Outcome at Day 14
Description: Description of clinical outcome in the Microbiological Intent-to-Treat (mITT) population. Responder (clinical outcome of improvement or response) was defined as survival with improvement or resolution of attributable signs and symptoms, and without new signs or symptoms, new foci of infection, change in antibiotics due to non-response, complications of S. aureus, or further surgery or medical intervention to treat S. aureus.
Time Frame: Day 14
Population: Microbiological Intent-to-Treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Responder (Improvement/Response) | 50 | 27
  Non-response | 18 | 13
  Indeterminate | 3 | 5
Statistical Analysis 1: Comparison: CF-301 vs Placebo; Test type: Other — Statistics considered descriptive as study designed to provide proof of concept and initial assessment of efficacy; not considered confirmatory; p = 0.3137, Fisher Exact; Risk Difference (RD) = 10.4, 90% CI 2-sided [-6.35 to 27.19]

3. Primary Outcome: CF-301 Maximum Plasma Concentration (Cmax)
Description: CF-301 plasma concentrations at specified timepoints.
Time Frame: Pre-dose and at 0.5, 1.5, 2, 2.25, 3, 4, 8, 14, 24, and 48 hours after the start of CF-301 infusion
Population: PK Population (patients with serial PK samples)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CF-301
Number analyzed (Participants) | 13
ng/mL | 1450.33 (636.83)

4. Primary Outcome: CF-301 Area Under the Curve (AUC 0-t)
Description: CF-301 plasma concentrations at specified time points
Time Frame: Pre-dose and at 0.5, 1.5, 2, 2.25, 3, 4, 8, 14, 24, and 48 hours after the start of CF-301 infusion
Population: PK Population (patients with serial PK samples)
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CF-301
Number analyzed (Participants) | 13
ng*hr/mL | 5667.42 (3032.03)

5. Secondary Outcome: Clinical Outcome at Day 7
Description: Description of clinical outcome in the mITT population. Responder (clinical outcome of improvement or response) was defined as survival with improvement or resolution of attributable signs and symptoms, and without new signs or symptoms, new foci of infection, change in antibiotics due to non-response, complications of S. aureus, or further surgery or medical intervention to treat S. aureus.
Time Frame: Day 7
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Responder (Improvement/Response) | 51 | 31
  Non-response | 17 | 11
  Indeterminate | 3 | 3

6. Secondary Outcome: Clinical Outcome at End of Standard of Care Antibacterial Therapy (EOT)
Description: as for outcome 5
Time Frame: EOT between 28-42 days
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Responder (Improvement/Response) | 44 | 28
  Non-response | 22 | 13
  Indeterminate | 5 | 4

7. Secondary Outcome: Clinical Outcome at Test of Cure (TOC)
Description: as for outcome 5
Time Frame: TOC between 56-70 days
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Responder (Improvement/Response) | 39 | 24
  Non-Response | 25 | 15
  Indeterminate | 7 | 6

8. Secondary Outcome: Clearance of Bacteremia at Day 7 After CF-301/Placebo Administration
Description: Number and percentage of patients with clearance of bacteremia in the mITT population
Time Frame: Day 7
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Clearance/presumed clearance of bacteremia | 59 | 39
  Ongoing bacteremia | 7 | 2
  Presumed ongoing bacteremia | 3 | 2
  Indeterminate | 2 | 2

9. Secondary Outcome: Clearance of Bacteremia at Day 14 After CF-301/Placebo Administration
Description: Number and percentage of patients with clearance of bacteremia in the mITT population
Time Frame: Day 14
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Clearance/presumed clearance of bacteremia | 64 | 38
  Ongoing bacteremia | 4 | 2
  Presumed ongoing bacteremia | 2 | 3
  Indeterminate | 1 | 2

10. Secondary Outcome: Microbiological Eradication at End of Standard of Care Antibacterial Therapy (EOT)
Description: Number and percentage of patients with microbiological eradication in the mITT population
Time Frame: EOT between 28-42 days
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Eradication/presumptive eradication | 50 | 31
  Persistence | 0 | 2
  Presumed persistence | 16 | 8
  Relapse | 0 | 0
  Indeterminate | 5 | 4

11. Secondary Outcome: Microbiological Eradication at Test of Cure (TOC)
Description: Number and percentage of patients with microbiological eradication in the mITT population
Time Frame: TOC between 56-70 days
Population: mITT population
Measure: Count of Participants; unit: Participants
Arm/Group | CF-301 | Placebo
Number analyzed (Participants) | 71 | 45
Participants
  Eradication/presumptive eradication | 46 | 31
  Persistence | 0 | 0
  Presumed persistence | 18 | 9
  Relapse | 0 | 0
  Indeterminate | 7 | 5

12. Other Pre Specified Outcome: Clinical Outcome at Day 14 in MRSA Subgroup
Description: Description of clinical outcome in the MRSA subgroup in the mITT population. Responder (clinical outcome of improvement or response) was defined as survival with improvement or resolution of attributable signs and symptoms, and without new signs or symptoms, new foci of infection, change in antibiotics due to non-response, complications of S. aureus, or further surgery or medical intervention to treat S. aureus.
Time Frame: Day 14
Population: Microbiological Intent-to-Treat (mITT) population
Measure: Count of Participants; unit: Participants
Groups:
- MRSA - CF-301: Patients in the MRSA Subgroup that received CF-301
- MRSA - Placebo: Patients in the MRSA Subgroup that received Placebo
Arm/Group | MRSA - CF-301 | MRSA - Placebo
Number analyzed (Participants) | 27 | 16
Participants
  Responder (Improvement/Response) | 20 | 5
  Non-response | 4 | 8
  Indeterminate | 3 | 3
Statistical Analysis 1: Comparison: MRSA - CF-301 vs MRSA - Placebo; Test type: Other — P-value was ad hoc. Statistics considered descriptive as study designed to provide proof of concept and initial assessment of efficacy; not considered confirmatory; p = 0.0101, Fisher Exact; Risk Difference (RD) = 42.8, 90% CI 2-sided [14.3 to 71.4]

13. Post Hoc Outcome: Clinical Responders at Day 14 in Patients With cBSI/R-IE
Description: Description of clinical responder at Day 14 in patients with complicated bloodstream infection (cBSI) / right-sided endocarditis (R-IE) (excluding left-sided endocarditis) in the mITT population. Responder (clinical outcome of improvement or response) was defined as survival with improvement or resolution of attributable signs and symptoms, and without new signs or symptoms, new foci of infection, change in antibiotics due to non-response, complications of S. aureus, or further surgery or medical intervention to treat S. aureus.
Time Frame: Day 14
Population: mITT population
Measure: Count of Participants; unit: Participants
Groups:
- cBSI/R-IE - CF-301: Patients with cBSI/R-IE that received CF-301
- cBSI/R-IE - Placebo: Patients with cBSI/R-IE that received Placebo
Arm/Group | cBSI/R-IE - CF-301 | cBSI/R-IE - Placebo
Number analyzed (Participants) | 47 | 39
Participants | 36 | 22
Statistical Analysis 1: Comparison: cBSI/R-IE - CF-301 vs cBSI/R-IE - Placebo; Test type: Other — P value was ad hoc. Descriptive statistics were performed; p = 0.0646, Fisher Exact; Descriptive statistics were performed

14. Post Hoc Outcome: Health Resource Utilization: Length of Hospital Stay
Description: Length of hospital stay in patients enrolled in the United States in the MRSA Subgroup in the mITT population
Time Frame: From study drug dosing to hospital discharge (in patients discharged alive) through Day 180
Population: Microbiological Intent-to-Treat (mITT) population
Measure: Median (Full Range); unit: days
Groups:
- MRSA, US - CF-301: Patients enrolled in the United States (discharged alive) in the MRSA Subgroup that received CF-301
- MRSA, US - Placebo: Patients enrolled in the United States (discharged alive) in the MRSA Subgroup that received Placebo
Arm/Group | MRSA, US - CF-301 | MRSA, US - Placebo
Number analyzed (Participants) | 25 | 13
days | 6 [2 to 69] | 10 [5 to 51]

15. Post Hoc Outcome: All-cause Mortality at Day 30 in MRSA Subgroup
Description: 30-day all-cause mortality in the MRSA subgroup in the mITT
Time Frame: Day 30
Population: Microbiological Intent-to-Treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | MRSA - CF-301 | MRSA - Placebo
Number analyzed (Participants) | 27 | 16
Participants | 1 | 4
Statistical Analysis 1: Comparison: MRSA - CF-301 vs MRSA - Placebo; Test type: Other — [test comment as in outcome 12, analysis 1]; p = 0.0556, Fisher Exact; Risk Difference (RD) = -21.3, 90% CI 2-sided [-45.1 to 2.5]

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected during the core study, from the time of consent through Test of Cure (TOC) between 56-70 days. After completion of the core study, all SAEs were collected during the long-term follow-up through Day 180.
Description: All-cause mortality is reported in the intent-to-treat (ITT) population. Serious adverse events and other (not including serious) adverse events are reported in the Safety population.
Arm/Group | CF-301 | Placebo
All-Cause Mortality (participants affected / at risk) | 17/73 | 9/48
Serious Adverse Events (participants affected / at risk) | 45/72 | 28/47
Other Adverse Events (participants affected / at risk) | 62/72 | 39/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CF-301 (N=72) | Placebo (N=47)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Splenic artery thrombosis (Blood and lymphatic system disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Impaired hearing (General disorders) | 1 | 0
Impaired self-care (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Arthritis bacterial (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 2 | 1
Staphylococcal bacteremia (Infections and infestations) | 2 | 3
Abscess bacterial (Infections and infestations) | 1 | 0
Arteriovenous graft site infection (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 2
Endocarditis (Infections and infestations) | 1 | 2
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Localized infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Necrotizing fasciitis (Infections and infestations) | 1 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Klebsiella bacteremia (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Septic embolus (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Ischemic cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Hemorrhage intracranial (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Procedure hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 1
Thrombosis in device (Product Issues) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Patient dissatisfaction with treatment (Social circumstances) | 0 | 1
Death NOS (General disorders) | 1 | 4 — Deaths recorded only on the Vital Status form were considered to have a fatal SAE of "death NOS", where NOS was not otherwise specified (for both the system organ class and preferred term).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CF-301 (N=72) | Placebo (N=47)
Anemia (Blood and lymphatic system disorders) | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Constipation (Gastrointestinal disorders) | 9 | 5
Diarrhea (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 6 | 3
Edema peripheral (General disorders) | 6 | 4
Pyrexia (General disorders) | 4 | 3
Cardiac murmur (Investigations) | 6 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 7 | 4
Anxiety (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 4 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 3
Hypotension (Vascular disorders) | 1 | 3
Urinary tract infection (Infections and infestations) | 8 | 6
Eye disorders (Ear and labyrinth disorders) | 5 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After multi-center publication has been published by sponsor, or if it hasn't been published in 24 months following completion of Clinical Study Report, PI may publish results independently. PI must allow sponsor at least 90 days to review submission, to request deletion of sponsor confidential information (not study results) and in that initial 90 day period, allow delay of up to 60 additional days to allow sponsor to protect its rights to any confidential information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03163446/Prot_SAP_000.pdf